CLINICAL TRIAL: NCT05851443
Title: A Phase 2, Double-Blind, Randomized, Placebo-Controlled, Dose-Ranging, Efficacy and Safety Study of Povorcitinib in Participants With Inadequately Controlled Moderate to Severe Asthma
Brief Title: A Study to Evaluate the Efficacy and Safety Study of Povorcitinib in Participants With Inadequately Controlled Moderate to Severe Asthma
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Incyte Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: INCB54707-208; 2022-502570-16-00 (Registry Identifier: EU CT Number)
Record Dates: First submitted 2023-04-24; First posted 2023-05-09 (Actual); Last update posted 2026-02-10 (Actual); Status verified 2026-02

CONDITIONS: Moderate to Severe Asthma
Keywords: Asthma; Moderate to Severe; INCB54707; Povorcitinib; ICS-LABA
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Inhaled Corticoseroid Long Acting Beta-Agonist(ICS-LABA) + placebo (Placebo Comparator): Participants will receive stable background therapy with ICS-LABA in combination with placebo once daily (QD) for 24 weeks during the placebo-controlled period. Participants will be allocated to 1 of 3 doses of povorcitinib during the extension period of 28 weeks
  Interventions: Other: placebo; Drug: ICS-LABA
- ICS-LABA + povorcitinib Dose 1 (Experimental): Participants will receive stable background therapy with ICS-LABA in combination with povorcitinib dose 1 once daily (QD) for 24 weeks during the placebo-controlled period, and Participants will continue to take the same dose of povorcitinib during the extension period of 28 weeks
  Interventions: Drug: povorcitinib; Drug: ICS-LABA
- ICS-LABA + povorcitinib Dose 2 (Experimental): Participants will receive stable background therapy with ICS-LABA in combination with povorcitinib dose 2 once daily (QD) for 24 weeks during the placebo-controlled period, and Participants will continue to take the same dose of povorcitinib during the extension period of 28 weeks
  Interventions: Drug: povorcitinib; Drug: ICS-LABA
- ICS-LABA + povorcitinib Dose 3 (Experimental): Participants will receive stable background therapy with ICS-LABA in combination with povorcitinib dose 3 once daily (QD) for 24 weeks during the placebo-controlled period, and Participants will continue to take the same dose of povorcitinib during the extension period of 28 weeks
  Interventions: Drug: povorcitinib; Drug: ICS-LABA

INTERVENTIONS:
Drug: povorcitinib — povorcitinib
  Other Names: INCB54707
  Arms: ICS-LABA + povorcitinib Dose 1; ICS-LABA + povorcitinib Dose 2; ICS-LABA + povorcitinib Dose 3
Other: placebo — placebo
  Arms: Inhaled Corticoseroid Long Acting Beta-Agonist(ICS-LABA) + placebo
Drug: ICS-LABA — Background Therapy

SUMMARY:
The study is being conducted to evaluate the effect of 3 dosing regimens of povorcitinib on pulmonary function

ELIGIBILITY:
Inclusion Criteria:

* Physician-diagnosed asthma requiring treatment with medium- to high-dose ICS-LABA for at least 12 months prior to screening.
* Pre-BD FEV1 < 80% predicted according to central over read value at Visit 2.
* Documented historical post-BD reversibility of FEV1 ≥ 12% and ≥ 200 mL in FEV1.
* At least 2 documented asthma exacerbations (requiring treatment with systemic CS, hospitalization, or emergency department visit) within 12 months prior to screening but not within the past 4 weeks prior to screening
* ACQ-6 ≥ 1.5 at screening.

Exclusion Criteria:

* Maintenance use of asthma controllers other than ICS-LABA.
* Have undergone bronchial thermoplasty.
* Current smokers or participants with a smoking history of ≥ 10 pack-years and participants using vaping products, including electronic cigarettes.
* Women who are pregnant (or who are considering pregnancy) or breastfeeding.
* Current conditions or history of other diseases, as follows:
* Clinically important pulmonary disease other than asthma ,Thrombocytopenia, coagulopathy, or platelet dysfunction.
* Venous and arterial thrombosis, deep vein thrombosis, pulmonary embolism, moderate to severe heart failure (NYHA Class III or IV), cerebrovascular accident, myocardial infarction, coronary stenting, or CABG surgery.
* Diagnosis of other significant cardiovascular diseases, including but not limited to angina, peripheral arterial disease, or uncontrolled arrhythmias such as atrial fibrillation, supraventricular tachycardia, ventricular tachycardia, and forms of carditis.
* Recipient of an organ transplant that requires continued immunosuppression.
* Immunocompromised (eg, lymphoma, acquired immunodeficiency syndrome, Wiskott-Aldrich syndrome).
* Any malignancies or history of malignancies.
* Chronic or recurrent infectious disease.
* Receipt of any biologic drugs used for asthma < 12 weeks or 5 half-lives (if known), whichever is longer, prior to screening

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 240 (Estimated)
Dates: Start 2023-07-11 (Actual); Primary Completion 2026-06-15 (Estimated); Study Completion 2027-01-31 (Estimated)

PRIMARY OUTCOMES:
Absolute change in pre-bronchodilator forced expiratory volume in the first 1 second (pre-BD FEV1) | Baseline ; Week 24
  To assess the effect of povorcitinib on lung function (pre-BD FEV1) between baseline and week 24

SECONDARY OUTCOMES:
Number of asthma exacerbations during the Placebo Controlled (PC) period | Up to 28 weeks
  Defined as a worsening of asthma
Absolute change from baseline in pre-BD FEV1 at each visit | Up to 14 months
Percent change from baseline in pre-BD FEV1 at each visit | Up to 14 months
Absolute change from baseline in post-BD FEV1 at week 24 | Baseline; Week 24
Percent change from baseline in post-BD FEV1 at week 24 | Baseline; Week 24
Absolute change from baseline in pre-BD FVC at each visit | Up to 14 months
Percent change from baseline in pre-BD FVC at each visit | Up to 14 months

CONTACTS AND LOCATIONS:
Locations (84):
- United States (26):
  - Allervie Clinical Research, Birmingham, Alabama
  - Kern Allergy Medical Clinic, Inc, Bakersfield, California
  - Integrated Research of Inland, Inc, Upland, California
  - Qway Research, Hialeah, Florida
  - Direct Helpers Research Center, Hialeah, Florida
  - Care Research Inc, Miami, Florida
  - Verus Clinical Research Corp, Miami, Florida
  - Dr. de Armas Research Center, Llc, Miami, Florida
  - Care Research Center, Inc, Miami, Florida
  - Anderson Allergy and Asthma, Orlando, Florida
  - Heuer Md Research Inc, Orlando, Florida
  - Advanced Clinical Research Atlanta, Atlanta, Georgia
  - Covenant Pulmonary Critical Care, East Point, Georgia
  - Northshore Medical Group, Glenview, Illinois
  - Henry Ford Hospital, Detroit, Michigan
  - Aa Medical Research Center, Flint, Michigan
  - Revive Research Institute, Southfield, Michigan
  - Northwell Health Physician Partners, New Hyde Park, New York
  - Pioneer Clinical Research Ny, New York, New York
  - Montefiore Medical Center (Mmc), The Bronx, New York
  - Onsite Clinical Solutions, Llc Charlotte Central Office, Charlotte, North Carolina
  - Temple University Hospital, Philadelphia, Pennsylvania
  - Clinical Research of Rock Hill, Rock Hill, South Carolina
  - Howland Allergy and Asthma Pllc Dba Orion Clinical Research, Austin, Texas
  - Linq Research, Llc, Pearland, Texas
  - Quality Assurance Research Center, San Antonio, Texas
- Argentina (23):
  - Fundacion Respirar, Buenos Aires
  - Fundacion Cidea, Buenos Aires
  - Mautalen Salud E Investigacion, Buenos Aires
  - INAER, Buenos Aires
  - Care: Centro de Alergia Y Enfermedades Respiratorias, CABA
  - Centro de Medicina Respiratoria, Concepción del Uruguay
  - Instituto de Medicina Respiratoria - Imer, Córdoba
  - CIMEL, Lanús
  - Fundacion Enfisema, Mar del Plata
  - Centro Medico Dharma, Mendoza
  - Polo de Salud Vistalba, Mendoza
  - Fundacion Scherbovsky, Mendoza
  - INSARES, Mendoza
  - Centro Respiratorio Quilmes, Quilmes
  - Centro Respiratorio Infantil, Rosario
  - Instituto de Diagnostico Abc, Rosario
  - Instituto Especialidades de La Salud Rosario, Rosario
  - Instituto Medico de La Fundacion Estudios Clinicos, Rosario
  - Centro Medico Respire, San Fernando
  - Ierim Instituto de Enfermedades Respiratorias E Investigacion Medica, San Juan Bautista
  - Ipr Instituto de Patologias Respiratorias, San Miguel de Tucumán
  - Cimer - Centro Integral de Medicina Respiratoria Srl, San Miguel de Tucumán
  - Iba Medica, Santa Fe
- Canada (6):
  - Synergy Respiratory Care, Sherwood Park, Alberta
  - Centre For Lung Health, Vancouver, British Columbia
  - Dynamic Drug Advancement, Ajax, Ontario
  - Ottawa Allergy Research Corporation, Ottawa, Ontario
  - S. Fikry Medicine Professional Corporation, Waterloo, Ontario
  - Dr. Syed Anees Medicine Professional Corporation, Windsor, Ontario
- Germany (5):
  - Pneumologische Gemeinschaftspraxis Kroker-Schaeben-Schmidt, Bendorf
  - Universitatsklinikum Bonn Aoer, Bonn
  - Ikf Pneumologie Frankfurt, Clinical Research Center Respiratory Diseases, Frankfurt am Main
  - Hannover Medical School, Hanover
  - Ikf Pneumologie Mainz, Mainz
- Japan (15):
  - Nihonbashi Medical and Allergy Clinic, Chūōku
  - Fukuwa Clinic, Chūōku
  - National Hospital Organization Fukuoka National Hospital, Fukuoka
  - Kishiwada City Hospital, Kishiwada
  - Kirigaoka Tsuda Hospital, Kitakyushu-shi
  - Tohno Chuo Clinic, Mizunami-shi
  - Kyosokai Amc Nishi-Umeda Clinic, Osaka
  - Lee Clinic, Osaka
  - Sakaide City Hospital, Sakaide-shi
  - Idaimae Minami Yojo Int Clinic, Sapporo
  - Tokyo Shinagawa Hospital, Shinagawa-ku
  - Takahashi Medical Clinic, Tokyo
  - Kouwa Clinic, Toshima-ku
  - Local Independent Administrative Institution Mie Prefectural General Medical Center, Yokkaichi-shi
  - Kaiseikai Kita Shin Yokohama Internal Medicine Clinic, Yokohama
- Poland (6):
  - Allergy Clinic Homeo Medicus, Bialystok
  - Uniwersyteckie Centrum Kliniczne, Gdansk
  - Nzoz Atopia, Krakow
  - Szpital Specjalistyczny Cdt Medicus, Lubin
  - Ostrowieckie Centrum Medyczne Spka Cywilna Anna Olech-Cudzik Krzysztof Cudzik, Ostrowiec Świętokrzyski
  - Pim Mswia, Warsaw
- Spain (3):
  - Giromed Institute/ Clinica Tres Torrres, Barcelona
  - Hospital Clinic Barcelona Main, Barcelona
  - Complejo Hospitalario Universitario de Santiago de Compostela, Santiago de Compostela

IPD SHARING:
Plan to Share IPD: Yes
Incyte shares data with qualified external researchers after a research proposal is submitted. These requests are reviewed and approved by a review panel on the basis of scientific merit. All data provided is anonymized to respect the privacy of patients who have participated in the trial in line with applicable laws and regulations. The trial data availability is according to the criteria and process described on https://www.incyte.com/our-company/compliance-and-transparency
Supporting Information: Study Protocol, SAP
Time Frame: Data will be shared after the primary publication or 2 years after the study has ended for market authorized products and indications.
Access Criteria: Data from eligible studies will be shared with qualified researchers according to the criteria and process described in the Data Sharing section of the www.incyteclinicaltrials.com website. For approved requests, the researchers will be granted access to anonymized data under the terms of a data sharing agreement.
URL: https://www.incyte.com/our-company/compliance-and-transparency

REFERENCES:
- See also: A Study to Evaluate the Efficacy and Safety Study of Povorcitinib in Participants With Inadequately Controlled Moderate to Severe Asthma — https://incyteclinicaltrials.com/studies/incb54707-208